CLINICAL TRIAL: NCT02470897
Title: A Phase I/II Study of Stereotactic Body Radiotherapy (SBRT) for Prostate Cancer Using Simultaneous Integrated Boost and Urethral-Sparing IMRT Planning
Brief Title: Stereotactic Body Radiation Therapy With Boost Using Urethral-Sparing Intensity-Modulated Radiation Therapy Planning in Treating Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW14083; NCI-2015-00950 (Registry Identifier: NCI Trial ID); 2015-0395 (Other: Institutional Review Board); UW14083 (Other: University of Wisconsin Carbone Cancer Center); A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison); Protocol Version 11/8/2023 (Other: UW Madison)
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stage I Prostate Adenocarcinoma; Stage II Prostate Adenocarcinoma
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (moderate dose SBRT with SIB) (Experimental): Patients undergo 5 fractions of moderate dose SBRT with SIB every other day for 10 days following urethral-sparing IMRT planning.
  SBRT: 8.0Gy escalated dose
  Interventions: Radiation: Radiation Therapy Treatment Planning and Simulation; Radiation: SBRT
- Arm B (uniform dose SBRT) (Active Comparator): Patients undergo 5 fractions of uniform dose SBRT every other day for 10 days following urethral-sparing IMRT planning.
  SBRT: 7.5Gy conventional dose
  Interventions: Radiation: Radiation Therapy Treatment Planning and Simulation; Radiation: SBRT

INTERVENTIONS:
Radiation: Radiation Therapy Treatment Planning and Simulation — Undergo urethral-sparing IMRT planning
  Other Names: Radiation Therapy Treatment Planning/Simulation
Radiation: SBRT — Undergo moderate dose SBRT with SIB
  Other Names: Stereotactic Body Radiation Therapy
  Arms: Arm A (moderate dose SBRT with SIB)
Radiation: SBRT — Undergo uniform dose SBRT
  Other Names: Stereotactic Body Radiation Therapy
  Arms: Arm B (uniform dose SBRT)

SUMMARY:
This phase I/II trial studies the side effects and best dose of stereotactic body radiation therapy while using intensity-modulated radiation therapy (IMRT) planning to help avoid radiation to normal tissue in patients with prostate cancer. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using small, high doses of radiation over several days and may cause less damage to normal tissue. This treatment schedule allows for a higher dose of radiation to be administered over a shorter overall treatment period in comparison to standard radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the incidence of genitourinary (GU) and gastrointestinal (GI) acute and late toxicity for patients treated with prostate stereotactic body radiotherapy (SBRT) with simultaneous integrative boost, urethral ring sparing, and enhanced prostate localization (magnetic resonance imaging [MRI\-computed tomography [CT] fusion).

II. To also evaluate the incidence of GU and GI acute and late toxicity for patients treated with prostate stereotactic body radiotherapy (SBRT) with a more conventional and uniformly delivered dose of 7.25 Gy/fraction to the prostate.

III. Disease-free survival: disease-free failure events include local progression, distant progression, biochemical failure as defined by the Radiation Therapy Oncology Group (RTOG) Phoenix definition, and death from any cause.

SECONDARY OBJECTIVES:

I. Evaluate patient quality of life (QOL) using the Expanded Prostate Cancer Index Composite 26 (EPIC-26) for evaluation of the QOL for up to 3 years after the completion of SBRT.

OUTLINE: Participants are assigned to 1 of 2 treatment arms. Participants unable to undergo MRI, whose MRI proves technically inadequate for delineating needed anatomic structures, or who decline to enroll on Arm A are assigned to Arm B.

ARM A: (n = 120) Participants undergo 5 fractions of moderate dose SBRT with simultaneous integrated boost (SIB) every other day for 10 days following urethral-sparing IMRT planning.

ARM B: (n = 40) Participants undergo 5 fractions of uniform dose SBRT every other day for 10 days following undergo urethral-sparing IMRT planning.

After completion of study treatment, patients are followed up at 4-8 weeks, at 4, 8, and 12 months, every 4 months for 1 year, every 6 months for 3 years, and then every 12 months thereafter.

Per protocol amendment in December 2023, the follow up time period for data collection will change to 3 years after the last participant completed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate and most recent biopsy within 180 days of study enrollment
* History/physical examination with digital rectal examination of the prostate within 90 days prior to study enrollment
* Gleason score =< 7, no tertiary pattern >= 5
* Clinical stage =< T2b (American Joint Committee on Cancer [AJCC] 7th Edition Staging Manual) and no radiographic evidence of T3 or T4 disease
* Clinical stage N0, M0
* Most recent prostate specific antigen (PSA) within 60 days of enrollment
* Maximum PSA =< 20 ng/ml (not within 20 days after biopsy)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* American Urological Association (AUA) =< 18 with or without medical management
* Up to a total of year of androgen deprivation allowed.
* Participant signs study specific informed consent prior to study enrollment

Exclusion Criteria:

* FOR ARM A: Inability to obtain a planning MRI or a planning MRI of sufficient quality to allow identification of the peripheral zone and urethra, or inability to adequately fuse the MRI to the planning CT scan
* FOR BOTH ARM A AND ARM B:
* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years; (for example, carcinoma in situ of the bladder or oral cavity is permissible)
* Prosthetic implants in the pelvic region that the investigator feels will impede treatment, planning, or delivery (e.g., an artificial hip)
* =< 3 months from a transurethral resection of the prostate (TURP) procedure
* Significant urinary obstruction (i.e. AUA symptom score > 18)
* Previous pelvic irradiation, prostate brachytherapy
* Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Severe, active comorbidity, defined as follows:

  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Crohn's disease or ulcerative colitis
  * Scleroderma

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Incidence of GU and GI Acute Toxicity | Up to 90 days
  Evaluation of delivering SBRT to the prostate using non-uniform dosing. The investigators will evaluate the potential for any added grade 3 rectal toxicity with the use of a simultaneous integrated boost.
Incidence of GU and GI Late Toxicity | Up to 3 years
  Evaluation of delivering SBRT to the prostate using non-uniform dosing. The investigators will evaluate the potential for any added grade 3 rectal toxicity with the use of a simultaneous integrated boost. A late adverse event will be defined as an adverse event occurring more than 90 days from the completion of RT.
Disease-free survival as measured by the Phoenix definition | Up to 3 years

SECONDARY OUTCOMES:
Change in Expanded Prostate Cancer Index Composite (EPIC) 26 Quality of Life Assessment | at Baseline, 1 year, and 2 years
  The EPIC 26 assessment has a total range of possible scores of 1-100 where higher scores indicate higher satisfaction. Questionnaires will be performed prior to treatment, and one and two years after completion of treatment.
Change in American Urological Association Symptom Score (AUASS) | at Baseline, 1 year, and 2 years
  The AUASS has a total possible range of scores of 0-35 where 1-7 is considered mild symptoms, 8-19 is considered moderate symptoms, and 20-35 is considered severe symptoms. Questionnaires will be performed prior to treatment, and one and two years after completion of treatment.
Change in International Index of Erectile Dysfunction Questionnaire (IIEF-5) | at Baseline, 1 year, and 2 years
  The IIEF-5 questionnaire has a total score of 1-25 where 1-7 is considered severe erectile dysfunction (ED), 8-11 is moderate ED, 12-16 is mild-moderate ED, 17-21 is mild ED, and 22-25 is no ED. Questionnaires will be performed prior to treatment, and one and two years after completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Morris, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Swedish American, Rockford, Illinois
  - UW Cancer Center, Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/